CLINICAL TRIAL: NCT00258622
Title: NS1209 and Lidocaine in Patients With Peripheral Neuropathic Pain: a Randomized, Double-Blind, Placebo-Controlled, Crossover Study
Brief Title: NS1209 and Lidocaine in Patients With Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Danish Pain Research Center (Other)
Collaborators: NeuroSearch A/S (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NS1209-008
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Pain
Keywords: Peripheral neuropathic pain; Neuropathic pain; Chronic pain
MeSH Terms: conditions — Pain; Neuralgia; Chronic Pain | interventions — SPD 502; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: NS1209
Drug: Lidocaine

SUMMARY:
Purpose: To evaluate the efficacy, tolerability and safety of NS1209 compared to lidocaine and placebo in patients with peripheral chronic neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Neuropathic pain and allodynia after a peripheral nerve injury (VAS >= 4)

Exclusion Criteria:

* Patients who cannot cooperate and do no understand Danish
* Fertile women
* Clinically significant abnormality or disease
* Drug and alcohol abuse
* Clinically abnormal ECG
* Hypersensitivity to any of the treatments
* Patients in treatment with cimetedin, antidepressants, antipsychotics, antiepileptics except gabapentin, anticoagulants, Na channel blockers and beta blockers
* Patients who have previously been treated in a NS1209 study
* Patients treated with an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-11; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
- Spontaneous ongoing pain intensity (VAS 0-100)

SECONDARY OUTCOMES:
Number of responders (at least 33% pain reduction)
Effect on evoked allodynia (VAS 0-100)
Pain relief for overall spontaneous pain (complete, good, moderate, slight, none or worse)
Feeling of unpleasantness (VAS 0-100)
Pain on movements (VAS 0-100)
Daily pain (NSP 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Troels S Jensen, MD, PhD, Principal Investigator — Danish Pain Research Center, Aarhus University Hospital
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark